CLINICAL TRIAL: NCT06732687
Title: Combined Effects of Calisthenics and Plyometric to Reduce Risk of Musculoskeletal Injuries Among School Going Children: A Randomized Clinical Trial
Brief Title: Combined Effects of Calisthenics and Plyometric to Reduce Risk of Musculoskeletal Injuries Among School Going Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RCRAHS-ISB/REC/MS-PT/01916
Record Dates: First submitted 2024-10-23; First posted 2024-12-13 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Musculoskeletal Injuries
Keywords: Risk of Musculoskeletal injuries; Calisthenics; Plyometrics; Combined ( Calisthenics + Plyometrics); Functional Movement Screening (FMS); Deep Squat; Shoulder mobility
MeSH Terms: interventions — Gymnastics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Calisthenics (Experimental): Experimental: Calisthenics Arm Description: Session will start with 9 minutes of warm up which includes 4 minutes of jogging and moderate intensity dynamic stretching for 5 minutes. Session would be of 8 minutes in which 1 minutes exercise and 1 minute rest is there. Exercise include bunny jumps, bear crawls , crab walk and mad cat and 9 minutes cool down period. This protocol would be follow up to 8 weeks.
  Interventions: Other: Calisthenics
- Plyometric (Experimental): Experimental: Plyometric
  Arm Description: Session will start with 9 minutes of warm up which includes 4 minutes of jogging and moderate intensity dynamic stretching for 5 minutes.. And 9 minutes cool down period. Following Plyometrics would be performed:1 medicine ball squats 2.ABC pushups 3.Medicine ball chest press 4.standing jump reach for star 5.SINGLE leg hops 6.Pushup on knees 7.zig zag double jump
  Interventions: Other: Plyometrics
- Combined( Calisthenics+ Plyometrics) (Experimental): Arm Description: In combined both calisthenics and plyometrics would be performed. First calisthenics will be performed and then plyometrics will be performed.
  Interventions: Other: Combined( Calisthenics+ Plyometrics)

INTERVENTIONS:
Other: Calisthenics — Calisthenics
  Arm Description: Session will start with 9 minutes of warm up which includes 4 minutes of jogging and moderate intensity dynamic stretching for 5 minutes. Session would be of 8 minutes in which 1 minutes exercise and 1 minute rest is there. Exercise include bunny jumps, bear crawls , crab walk and mad cat and 9 minutes cool down period. This protocol would be follow up to 8 weeks.
  Arms: Calisthenics
Other: Plyometrics — Description: Session will start with 9 minutes of warm up which includes 4 minutes of jogging and moderate intensity dynamic stretching for 5 minutes.. And 9 minutes cool down period. Following Plyometrics would be performed:1 medicine ball squats 2.ABC pushups 3.Medicine ball chest press 4.standing jump reach for star 5.SINGLE leg hops 6.Pushup on knees 7.zig zag double jump
  Arms: Plyometric
Other: Combined( Calisthenics+ Plyometrics) — Description: Both exercises would be performed. First Calisthenics will be performed and then plyometrics will be performed.
  Arms: Combined( Calisthenics+ Plyometrics)

SUMMARY:
The goal of this clinical trial is to know about the combined effects of calisthenics and plyometric exercises on reducing risk of MSK injuries among school-going children. The main questions it aims to answer are:

1. Will combined exercises (calisthenics+ plyometrics) have a better effect on reducing risk of MSK injuries among school-going children?
2. How do these exercise interventions impact functional movements, and musculoskeletal pain improvements in children Researchers will compare a calisthenics exercise group, a plyometric exercise group, and a combined group (Calisthenics+ Plyometric) to see if there are differences in reducing risk of MSK injuries outcomes.

Participants will:

* Be male school-going children aged 8-12 years.
* Be randomly assigned to one of three groups: calisthenics, plyometric, or combined
* Complete baseline assessments of MSK (Functional Movement Screening and pain).
* Participate in their assigned exercise program 3 times per week for 8 weeks
* Complete follow-up assessments of MSK (Functional Movement Screening and pain) at 4 weeks and 8 weeks.
* Perform tests for functional movement screening and MSK assessment.

DETAILED DESCRIPTION:
Title: Combined effects of Calisthenics and Plyometric Exercises on reducing risk of MSK Injuries Among School-Going Children.

This research study, conducted by Adeeba Tabassum at Riphah International University in Islamabad, aims to investigate how different types of exercise can reduce MSK injuries in children. Specifically, it tell us the effects of combined (calisthenics+ plyometrics), calisthenics (bodyweight exercises) , plyometrics (jump training) on reducing risk of MSK Injuries in school-going children.

Key Details:

* Participants: Male school-going children aged 8-12 years
* Duration: 8 weeks
* Location: Public and private schools in Islamabad, Pakistan

The study will involve three groups:

1. Calisthenics group: Performing bodyweight exercises
2. Plyometric group: Engaging in jumping and explosive movement exercises
3. Combined group: Calisthenics+ Plyometric Calisthenics group will participate in supervised sessions three times per week and plyometric and combined will 2 times per week. The exercises are designed to be age-appropriate and safe for children.

Measurements:

Researchers will assess various aspects of MSK function using standardized tests:

- TNMQ'S FMS These assessments will be conducted at the beginning of the study, at 4 weeks, and at 8 weeks to track changes over time.

Significance:

This study is important because it could provide valuable insights into how different types of exercise reduces risk of MSK Injuries. The results could inform physical education programs in schools and help parents and educators make informed decisions about children's physical activities.

Ethical Considerations:

The study has been approved by the university's ethics review board. Participation is voluntary, and parents must provide informed consent. All data will be kept confidential and coded to protect participants' identities.

Expected Outcomes:

The researchers hypothesize that calisthenics exercises may have a more significant positive effect on reducing risk of MSK Injuries compared to plyometric exercises. However, both exercise types are expected to show improvements compared to the control group.

This research contributes to the growing field of exercise neuroscience and could have practical implications for child development, education, and public health policies related to physical activity in schools.

ELIGIBILITY:
Inclusion Criteria:

* Male School Going Children (8-12 Years Of Age)
* Normal BMI of School Going Children
* No Recent Musculoskeletal Injury from last month.
* Not Actively Engaged In Other Sports

Exclusion Criteria:

* Children with any mental or physical disability.
* Children with acute illness or fracture
* Active Inflammation or infections
* Any physical deformity

Ages: 8 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Male participant are included in the study
Enrollment: 99 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-04-04 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
DEEP SQUAT Test (Functional movement screening) | 8 weeks
  The Deep Squat Test is a key component of the Functional Movement Screen (FMS) used to assess an individual's overall mobility, stability, and movement patterns.
  In this test, the 33 participants are asked to perform a deep squat with their feet shoulder-width apart, toes pointing forward, and arms extended overhead. The goal is to squat as deeply as possible while maintaining proper form, including a neutral spine, stable knees, and balanced feet.
  Sets/Repetitions: 2/8
Hurdle step Test (Functional movement screening) | 8 weeks
  The Hurdle Step Test is part of the Functional Movement Screen (FMS), a tool used to assess movement patterns and identify potential areas of dysfunction or risk for injury.
  In this test, the individual is required to step over a hurdle while maintaining a controlled stance. The hurdle is typically set at a height that challenges the individual's flexibility, mobility, and stability. The movement is performed while focusing on proper alignment and balance.
INCLINE LUNGES Test (Functional movement screening) | 8 weeks
  The Incline Lunges Test is a component of functional movement screening designed to evaluate an individual's lower body strength, stability, and mobility. It specifically assesses the coordination between the hip, knee, and ankle joints while testing the flexibility of the hip flexors and the stability of the core and pelvis.
Shoulder Mobility Test Functional movement screening (FMS) | 8 weeks
  To do this test, stand up straight and make a fist with each hand. Place one fist on opposite shoulder and the other behind back on the same side. Try to bring elbows as close as possible without moving torso.
Impingement clearing test (Functional movement screening (FMS) | 8 weeks
  The shoulder clearing test is a pain-free procedure that checks for shoulder impingement:
  Reach hand across body and place it against opposite shoulder. Apply inward pressure while slowly raising elbow. Repeat on the other side.
Active straight leg raise (Functional movement screening (FMS) | 8 weeks
  The subject is instructed to raise one leg, then the other, without bending the knee, until the heel is 20 cm above the table.
  The subject is asked to hold the leg elevated for about 10 seconds. The subject is asked to rate the difficulty of the test on a scale of 0 to 5. The subject is asked if one leg feels heavier than the other or if there is any pain.
Trunk stability pushups (Functional movement screening (FMS) | 8 weeks
  Lie on stomach with hands shoulder-width apart Position thumbs in line with forehead if male, or chin if female Tighten core and raise body off the ground in one line Try to arch back as little as possible Push body up into a push-up position as one unit Ensure there's no lag in spine
Press up clearing test (Functional movement screening (FMS) | 8 weeks
  The press-up clearing test is a part of the Functional Movement Screen (FMS) that assesses pain response and is used to identify individuals at risk of injury:
  Position The participant lies on their stomach with their hands placed shoulder-width apart and palms down.
  Instructions The participant should raise their toes toward their shins and place them on the ground, extend their knees, and maintain a rigid torso.
  Execution The participant should press their chest off the floor by extending their elbows, arching their back as much as possible, and keeping their hips in contact with the floor.
  Scoring If the participant experiences pain at any point during the test, receive a score of zero and the test is terminated. The painful area should be noted.
Rotary stability (Functional movement screening (FMS) | 8 weeks
  The procedure involves the following steps:
  Get on all fours with hands and knees on a board, with arms and thighs vertical and toes resting on the floor.
  Simultaneously reach right arm forward and extend right leg backward. Retract elbow and right knee until touch directly over the board. Repeat the movement at least twice without touching the floor with arm or leg. Repeat the test on the other side. If you can't complete the movement within three attempts, you can try a modified diagonal flexion and extension lift.
  The test administrator will assess performance based on whether hand and leg clear the floor by about 6 inches (15 cm) and whether you make contact with the floor while performing the repetitions
Posterior Rocking Clearing Test (Functional Movement Screening (FMS) | 8 weeks
  Posterior rocking clearing test is performed:
  Assume a quadruped position Rock back and touch the buttocks to the heels and the chest to the thighs Keep the hands in front of the body and reach out as far as possible
  The FMS is a series of seven tests that evaluate fundamental movement patterns. The tests are designed to identify movements that increase the risk of injury and insufficient movement that reduces performance. The FMS uses a four-point scale to score each test:
  3: The movement task was performed perfectly without compensations 2: The task was completed with compensatory movements
  1: The participant was unable to perform the movement as required 0: The participant felt pain during the movement task

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmed Awan, PHD, Principal Investigator — Riphah International University
Locations (1):
- Different Schools, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No